CLINICAL TRIAL: NCT01388673
Title: Open Prospective Study to Evaluate the Safety and Preliminary Effectiveness of the BaroSense ACE Stapler for Plication of Dilated Post-surgical Gastric Anatomy
Brief Title: Safety and Preliminary Effectiveness of the BaroSense Articulating Circular Endoscopic (ACE) Stapler for Plication of Dilated Post-surgical Gastric Anatomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: BaroSense Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 11-02
Record Dates: First submitted 2011-07-01; First posted 2011-07-07 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Obese
Keywords: prior RYGB procedure; regained weight over time; dilated pouch and/or stoma
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACE Stapler procedure (Experimental): ACE Stapler procedure for the treatment of dilated post-surgical gastric anatomy
  Interventions: Procedure: BaroSense ACE Stapler for plication of dilated post-surgical gastric anatomy

INTERVENTIONS:
Procedure: BaroSense ACE Stapler for plication of dilated post-surgical gastric anatomy — The ACE Stapler is used endoscopically, an incorporates a unique tissue capture mechanism to produce large, permanent serosa to serosa plications in a completely trans-oral approach.

SUMMARY:
The BaroSense Articulating Circular Endoscopic (ACE) Stapler is an investigational instrument indicated for endoluminal trans-oral tissue approximation and ligation in the gastrointestinal tract. This study explores the specific application of tissue apposition in dilated post-surgical gastric anatomy such as observed in a dilated Roux-en-Y Gastric Bypass (RYGB) pouch.

The primary objective of this study is to perform an evaluation of the safety of the ACE Stapler for the treatment of dilated post-surgical gastric anatomy.

The secondary objective of this study is to evaluate the preliminary efficacy of the ACE Stapler for the treatment of dilated post-surgical gastric anatomy over a 12 month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject, male or female, is age 18 to 60 years of age.
2. Subject must be able to understand and be willing to sign an informed consent document.
3. Subject must be willing and able to participate in all aspects of the study and agree to comply with all study requirements for the duration of the study. This includes availability of reliable transportation and sufficient time to attend all follow-up visits.
4. Subject must be > 2 years post RYGB surgery.
5. Subject must have documented records indicating an initial achievement of > 60% EWL (based on an ideal weight of 25 BMI) at some point after RYGB surgery.
6. Subject has a BMI at baseline of > 30 and < 50.
7. At time of enrollment, subject must have regained at least 35% of the maximum weight lost following RYGB, and the weight regain must have occurred over a period of not less than 3 months from the point of maximum weight loss.
8. Subject must have a stoma diameter of at least 18 mm.
9. Subject must be fully ambulatory, without chronic reliance on walking aids such as crutches, walkers or a wheelchair.

Exclusion Criteria:

1. Subject has a severe eating disorder.
2. Investigator determines that there is another causal factor for the subject's weight regain other than dilated gastric anatomy.
3. Subject has previously undergone an endoscopic or surgical repair of dilated pouch or stoma (including sclerotherapy treatments).
4. Subject had irreversible or life threatening complications following initial RYGB procedure (cardio or respiratory).
5. Subject has an ongoing severe complication from their initial RYGB procedure (recurrent ventral hernia, pain syndrome, etc.).
6. Subject has an intragastric fistula, anastomotic leak, or staple/suture line disruption.
7. Subject has history of/or signs and/or symptoms of gastro-duodenal ulcer disease.
8. Subject has symptomatic congestive heart failure, cardiac arrhythmia or unstable coronary artery disease.
9. Subject has pre-existing respiratory disease such as chronic obstructive pulmonary disease (COPD), pneumonia or cancer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with adverse events | Post-procedure through 12 months
  The primary safety analysis will assess the occurrence of adverse events through 12 months following procedures. Included in this assessment will be the proportion of subjects with any of the following outcomes between enrollment and completion of the 12 month follow-up evaluation: Adverse Events (AE), Adverse Device Effects (ADE), Serious Adverse Events (SAE) and Unanticipated Adverse Device Effects (UADE).

SECONDARY OUTCOMES:
Percent excess weight loss in participants relative to preop weight | Through 12 months post-procedure
  Efficacy measurements will be analyzed relative to the surgery visit. The collected measures will include:
  * Percent Excess Weight Loss (%EWL) defined as: (preop weight-current weight)/ (preop weight - ideal weight) *100, where ideal weight is calculated from a BMI of 25 based on the subject's height.
  * Total weight lost (kg)
  * Change in body mass index (BMI)
  * Change in waist circumference
  * Improvement in co-morbid disease(s) including, but not limited to, improvement in vital signs and/or laboratory values